CLINICAL TRIAL: NCT02300753
Title: Emergency Administration of EPI-743 to a Single Patient With Leber's Hereditary Optic Neuropathy [LHON]
Status: No longer available | Type: Expanded Access
Sponsor: Edison Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: EPI-2010-004
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Leber's Hereditary Optic Neuropathy
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — alpha-tocotrienol quinone

INTERVENTIONS:
Drug: EPI-743 — EPI-743 is a quinone oxidation product of alpha-tocotrienol
  Other Names: Vincerinone (TM); Vatiquinone

SUMMARY:
Expanded access Protocol to treat LHON subjects with EPI743

DETAILED DESCRIPTION:
Emergency use administration of EPI-743 to subjects with LHON. This Protocol was originally developed to treat a single subject but was expanded to treat several at a single institution.

ELIGIBILITY:
Inclusion Criteria:

* Emergency treatment for subjects with LHON who are actively losing site in one eye

Exclusion Criteria:

* Allergy to EPI-743 or sesame oil
* Clinical history of bleeding or abnormal PT/PTT
* Hepatic insufficiency with LFTs greater than 2-times normal
* Renal insufficiency requiring dialysis
* Fat malabsorption syndromes
* Any other concurrent inborn erros of metabolism
* Severe end-organ hypo-perfusion syndrome secondary to cardiac failure resulting in lactic acidosis
* Anemia with a HCT <25

Ages: 8 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Doheny Eye Institute / UCLA, Los Angeles, California, United States